CLINICAL TRIAL: NCT04508985
Title: Management of Renin-Angiotensin-Aldosterone System Blockade in Patients Admitted in Hospital With Confirmed Coronavirus Disease (COVID-19) Infection: The McGill RAAS-COVID-19 Randomized Controlled Trial
Brief Title: The McGill RAAS-COVID-19 Trial
Acronym: RAAS-COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Jewish General Hospital (Montreal, Quebec, Canada) (Unknown); Montreal General Hospital (Montreal, Quebec, Canada) (Unknown); Université de Lorraine, Centre d'Investigation Clinique- Plurithématique Inserm (Unknown)
Responsible Party: Principal Investigator, Abhinav Sharma, Cardiologist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MP-37-2021-6614
Record Dates: First submitted 2020-08-10; First posted 2020-08-11 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: COVID-19; Cardiovascular Diseases
Keywords: Renin; Angiotensin; Aldosterone; coronavirus; Cardiovascular Diseases; COVID-19
MeSH Terms: conditions — COVID-19; Cardiovascular Diseases; Coronavirus Infections | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Open-label, randomized, study of approximately 40 adults. The following groups of participants will be considered: i) within 48 hours of diagnosis of COVID-19; ii) who have received a diagnosis of COVID-19 from another facility and are within 48 hours of transfer to a study recruitment site (Royal Victoria Hospital, Montreal General Hospital, and Jewish General Hospital [all in Montreal, Quebec, Canada])). Participants will be randomized 1:1 to an upfront temporary discontinuation) of RAAS inhibition for the duration of the hospitalization (and to consider re-initiate on discharge) versus a strategy continuation of RAAS inhibition.
Masking Description: The patient and the treating doctor will be informed of the assigned treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Temporarily holding the RAAS inhibitor. Among participants who will be randomized to the intervention arm, a possible guideline-directed alternative to anti-hypertensive medication alternatives will be provided to the treating physician team.
  Interventions: Other: Temporarily holding the RAAS inhibitor [intervention]
- Continuation of standard of care (Other): No intervention, Continuation RAAS inhibitor [continued standard of care].
  Interventions: Other: RAAS inhibitor [continued standard of care]

INTERVENTIONS:
Other: Temporarily holding the RAAS inhibitor [intervention] — Temporarily holding the RAAS inhibitor. Among participants who will be randomized to the intervention arm, a possible guideline-directed alternative to anti-hypertensive medication alternatives will be provided to the treating physician team.
  Arms: Intervention
Other: RAAS inhibitor [continued standard of care] — No intervention, Continuation RAAS inhibitor [continued standard of care].
  Arms: Continuation of standard of care

SUMMARY:
Coronavirus disease (COVID-19) related pneumonia significantly impact patients with underlying cardiovascular (CV) conditions. Animal studies suggest that drugs commonly used to treated CV diseases may increase the ability of COVID-19 to infect cells. The RAAS-COVID-19 trial aims to assess whether temporarily holding these CV drugs in patients who are admitted with COVID-19, versus continuing them, in patients admitted with COVID-19 can impact short term outcomes.

DETAILED DESCRIPTION:
Open-label, pragmatic, randomized, study of approximately 40 adults. The following groups of participants will be considered: i) within 48 hours of diagnosis of COVID-19; ii) who have received a diagnosis of COVID-19 from another facility and are within 48 hours of transfer to a study recruitment site (Royal Victoria Hospital, Montreal General Hospital, and Jewish General Hospital [all in Montreal, Quebec, Canada]). Participants will be randomized 1:1 to an upfront temporary discontinuation) of RAAS inhibition for the duration of the hospitalization (and to consider re-initiate after day 7 of admission or on discharge) versus a strategy continuation of RAAS inhibition. Re-initiation of held RAAS inhibition will be based on treating team's clinical judgement. The RAAS-COVID-19 RCT will evaluate whether an upfront strategy of temporary discontinuation of RAAS inhibition compared to the continuation of RAAS inhibition among patients admitted with established COVID-19 infection and on chronic RAAS inhibition therapy impacts short term clinical outcomes and biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Hospitalization with a Covid-19 infection
* Chronically treated with RAAS blockers (ACE inhibitors or ARBs on the last prescription prior to admission with a treatment duration ≥ 1 month
* Diagnosis of COVID-19 confirmed by the presence of SARS-CoV-2 on any biological sample
* Participants are within 48 hours of diagnosis of COVID-19 or have received a diagnosis of COVID-19 from another facility and are within 48 hours of transfer to a study recruitment site

Exclusion Criteria:

* Shock requiring vasoactive agents.
* Requiring invasive mechanical ventilation.
* History of malignant hypertension
* Use of five or more antihypertensive drugs.
* History of heart failure with reduced ejection fraction
* History of hospitalization for acute heart failure in past 3 months
* History of hospitalization for hemorrhagic stroke in the past 3 months.
* History of CKD with an eGFR <45 ml/min/1.73m2
* History of COPD GOLD III/IV
* History of end-stage dementia
* History of active liver cirrhosis
* RAAS blockers therapy previously stopped > 48h.
* Anticipated discharge in less than 24 hours.
* History of current active cancer receiving chemotherapy
* Inability to obtain informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-17 (Actual)

PRIMARY OUTCOMES:
Global rank score | Baseline - day 7
  The primary end point is a global rank score which is applied to all participants. The global rank sum is based on the following endpoints (and corresponding score): Death (7); Transfer to ICU for Invasive ventilation (6); Transfer to ICU for other indication (5); Non-fatal MACE (Any of the following - MI, Stroke, Acute HF, new onset Afib) (4); Length of stay > 4 days (3); Development of acute kidney injury (>40% decline in eGFR or doubling of serum Cr) (2); Urgent intravenous treatment for high blood pressure/hypertensive crisis (2); >30% Increase in baseline high sensitivity troponin (1); >30% increase in baseline BNP (1); Increase in baseline CRP to 48 hours >30%(1); Lymphocyte count drop >30% (1).
  The primary endpoint will be assessed from baseline to day 7 (or day of discharge if occurs before day 7). Participants will receive a weighted score depending on the events experienced. The global rank sum score will then be averaged and compared between treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Abhinav Sharma, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Muhc-Rimuhc, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data will be de-identified and shared among all collaborators.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediate access to the data

REFERENCES:
- [Background] Brown PM, Ezekowitz JA. Composite End Points in Clinical Trials of Heart Failure Therapy: How Do We Measure the Effect Size? Circ Heart Fail. 2017 Jan;10(1):e003222. doi: 10.1161/CIRCHEARTFAILURE.116.003222. PMID 28077429
- [Background] Kuhn JH, Li W, Choe H, Farzan M. Angiotensin-converting enzyme 2: a functional receptor for SARS coronavirus. Cell Mol Life Sci. 2004 Nov;61(21):2738-43. doi: 10.1007/s00018-004-4242-5. PMID 15549175
- [Background] Ferrario CM, Jessup J, Chappell MC, Averill DB, Brosnihan KB, Tallant EA, Diz DI, Gallagher PE. Effect of angiotensin-converting enzyme inhibition and angiotensin II receptor blockers on cardiac angiotensin-converting enzyme 2. Circulation. 2005 May 24;111(20):2605-10. doi: 10.1161/CIRCULATIONAHA.104.510461. Epub 2005 May 16. PMID 15897343
- [Background] Agata J, Ura N, Yoshida H, Shinshi Y, Sasaki H, Hyakkoku M, Taniguchi S, Shimamoto K. Olmesartan is an angiotensin II receptor blocker with an inhibitory effect on angiotensin-converting enzyme. Hypertens Res. 2006 Nov;29(11):865-74. doi: 10.1291/hypres.29.865. PMID 17345786
- [Background] Kuster GM, Pfister O, Burkard T, Zhou Q, Twerenbold R, Haaf P, Widmer AF, Osswald S. SARS-CoV2: should inhibitors of the renin-angiotensin system be withdrawn in patients with COVID-19? Eur Heart J. 2020 May 14;41(19):1801-1803. doi: 10.1093/eurheartj/ehaa235. No abstract available. PMID 32196087
- [Background] Sharma A, Bhatt DL, Calvo G, Brown NJ, Zannad F, Mentz RJ. Heart failure event definitions in drug trials in patients with type 2 diabetes. Lancet Diabetes Endocrinol. 2016 Apr;4(4):294-6. doi: 10.1016/S2213-8587(16)00049-8. No abstract available. PMID 27016320
- [Background] Marquis-Gravel G, Roe MT, Turakhia MP, Boden W, Temple R, Sharma A, Hirshberg B, Slater P, Craft N, Stockbridge N, McDowell B, Waldstreicher J, Bourla A, Bansilal S, Wong JL, Meunier C, Kassahun H, Coran P, Bataille L, Patrick-Lake B, Hirsch B, Reites J, Mehta R, Muse ED, Chandross KJ, Silverstein JC, Silcox C, Overhage JM, Califf RM, Peterson ED. Technology-Enabled Clinical Trials: Transforming Medical Evidence Generation. Circulation. 2019 Oct 22;140(17):1426-1436. doi: 10.1161/CIRCULATIONAHA.119.040798. Epub 2019 Oct 21. PMID 31634011
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Arentz M, Yim E, Klaff L, Lokhandwala S, Riedo FX, Chong M, Lee M. Characteristics and Outcomes of 21 Critically Ill Patients With COVID-19 in Washington State. JAMA. 2020 Apr 28;323(16):1612-1614. doi: 10.1001/jama.2020.4326. PMID 32191259
- [Background] Ye M, Wysocki J, William J, Soler MJ, Cokic I, Batlle D. Glomerular localization and expression of Angiotensin-converting enzyme 2 and Angiotensin-converting enzyme: implications for albuminuria in diabetes. J Am Soc Nephrol. 2006 Nov;17(11):3067-75. doi: 10.1681/ASN.2006050423. Epub 2006 Oct 4. PMID 17021266
- [Background] Soler MJ, Ye M, Wysocki J, William J, Lloveras J, Batlle D. Localization of ACE2 in the renal vasculature: amplification by angiotensin II type 1 receptor blockade using telmisartan. Am J Physiol Renal Physiol. 2009 Feb;296(2):F398-405. doi: 10.1152/ajprenal.90488.2008. Epub 2008 Nov 12. PMID 19004932
- [Background] Vuille-dit-Bille RN, Camargo SM, Emmenegger L, Sasse T, Kummer E, Jando J, Hamie QM, Meier CF, Hunziker S, Forras-Kaufmann Z, Kuyumcu S, Fox M, Schwizer W, Fried M, Lindenmeyer M, Gotze O, Verrey F. Human intestine luminal ACE2 and amino acid transporter expression increased by ACE-inhibitors. Amino Acids. 2015 Apr;47(4):693-705. doi: 10.1007/s00726-014-1889-6. Epub 2014 Dec 23. PMID 25534429
- [Background] Vaduganathan M, Vardeny O, Michel T, McMurray JJV, Pfeffer MA, Solomon SD. Renin-Angiotensin-Aldosterone System Inhibitors in Patients with Covid-19. N Engl J Med. 2020 Apr 23;382(17):1653-1659. doi: 10.1056/NEJMsr2005760. Epub 2020 Mar 30. No abstract available. PMID 32227760
- [Background] Bavishi C, Maddox TM, Messerli FH. Coronavirus Disease 2019 (COVID-19) Infection and Renin Angiotensin System Blockers. JAMA Cardiol. 2020 Jul 1;5(7):745-747. doi: 10.1001/jamacardio.2020.1282. No abstract available. PMID 32242890
- [Background] Zhang P, Zhu L, Cai J, Lei F, Qin JJ, Xie J, Liu YM, Zhao YC, Huang X, Lin L, Xia M, Chen MM, Cheng X, Zhang X, Guo D, Peng Y, Ji YX, Chen J, She ZG, Wang Y, Xu Q, Tan R, Wang H, Lin J, Luo P, Fu S, Cai H, Ye P, Xiao B, Mao W, Liu L, Yan Y, Liu M, Chen M, Zhang XJ, Wang X, Touyz RM, Xia J, Zhang BH, Huang X, Yuan Y, Loomba R, Liu PP, Li H. Association of Inpatient Use of Angiotensin-Converting Enzyme Inhibitors and Angiotensin II Receptor Blockers With Mortality Among Patients With Hypertension Hospitalized With COVID-19. Circ Res. 2020 Jun 5;126(12):1671-1681. doi: 10.1161/CIRCRESAHA.120.317134. Epub 2020 Apr 17. PMID 32302265
- [Background] Guo J, Huang Z, Lin L, Lv J. Coronavirus Disease 2019 (COVID-19) and Cardiovascular Disease: A Viewpoint on the Potential Influence of Angiotensin-Converting Enzyme Inhibitors/Angiotensin Receptor Blockers on Onset and Severity of Severe Acute Respiratory Syndrome Coronavirus 2 Infection. J Am Heart Assoc. 2020 Apr 7;9(7):e016219. doi: 10.1161/JAHA.120.016219. Epub 2020 Apr 1. No abstract available. PMID 32233755
- [Background] Sun H, Davison BA, Cotter G, Pencina MJ, Koch GG. Evaluating treatment efficacy by multiple end points in phase II acute heart failure clinical trials: analyzing data using a global method. Circ Heart Fail. 2012 Nov;5(6):742-9. doi: 10.1161/CIRCHEARTFAILURE.112.969154. Epub 2012 Oct 11. PMID 23065036
- [Background] Felker GM, Maisel AS. A global rank end point for clinical trials in acute heart failure. Circ Heart Fail. 2010 Sep;3(5):643-6. doi: 10.1161/CIRCHEARTFAILURE.109.926030. No abstract available. PMID 20841546
- [Background] Margulies KB, Hernandez AF, Redfield MM, Givertz MM, Oliveira GH, Cole R, Mann DL, Whellan DJ, Kiernan MS, Felker GM, McNulty SE, Anstrom KJ, Shah MR, Braunwald E, Cappola TP; NHLBI Heart Failure Clinical Research Network. Effects of Liraglutide on Clinical Stability Among Patients With Advanced Heart Failure and Reduced Ejection Fraction: A Randomized Clinical Trial. JAMA. 2016 Aug 2;316(5):500-8. doi: 10.1001/jama.2016.10260. PMID 27483064
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Sharma A, Hijazi Z, Andersson U, Al-Khatib SM, Lopes RD, Alexander JH, Held C, Hylek EM, Leonardi S, Hanna M, Ezekowitz JA, Siegbahn A, Granger CB, Wallentin L. Use of Biomarkers to Predict Specific Causes of Death in Patients With Atrial Fibrillation. Circulation. 2018 Oct 16;138(16):1666-1676. doi: 10.1161/CIRCULATIONAHA.118.034125. PMID 29871978
- [Background] Clerkin KJ, Fried JA, Raikhelkar J, Sayer G, Griffin JM, Masoumi A, Jain SS, Burkhoff D, Kumaraiah D, Rabbani L, Schwartz A, Uriel N. COVID-19 and Cardiovascular Disease. Circulation. 2020 May 19;141(20):1648-1655. doi: 10.1161/CIRCULATIONAHA.120.046941. Epub 2020 Mar 21. PMID 32200663
- [Background] Nerenberg KA, Zarnke KB, Leung AA, Dasgupta K, Butalia S, McBrien K, Harris KC, Nakhla M, Cloutier L, Gelfer M, Lamarre-Cliche M, Milot A, Bolli P, Tremblay G, McLean D, Padwal RS, Tran KC, Grover S, Rabkin SW, Moe GW, Howlett JG, Lindsay P, Hill MD, Sharma M, Field T, Wein TH, Shoamanesh A, Dresser GK, Hamet P, Herman RJ, Burgess E, Gryn SE, Gregoire JC, Lewanczuk R, Poirier L, Campbell TS, Feldman RD, Lavoie KL, Tsuyuki RT, Honos G, Prebtani APH, Kline G, Schiffrin EL, Don-Wauchope A, Tobe SW, Gilbert RE, Leiter LA, Jones C, Woo V, Hegele RA, Selby P, Pipe A, McFarlane PA, Oh P, Gupta M, Bacon SL, Kaczorowski J, Trudeau L, Campbell NRC, Hiremath S, Roerecke M, Arcand J, Ruzicka M, Prasad GVR, Vallee M, Edwards C, Sivapalan P, Penner SB, Fournier A, Benoit G, Feber J, Dionne J, Magee LA, Logan AG, Cote AM, Rey E, Firoz T, Kuyper LM, Gabor JY, Townsend RR, Rabi DM, Daskalopoulou SS; Hypertension Canada. Hypertension Canada's 2018 Guidelines for Diagnosis, Risk Assessment, Prevention, and Treatment of Hypertension in Adults and Children. Can J Cardiol. 2018 May;34(5):506-525. doi: 10.1016/j.cjca.2018.02.022. Epub 2018 Mar 1. PMID 29731013
- [Derived] Sharma A, Elharram M, Afilalo J, Flannery A, Afilalo M, Tselios C, Ni J, Ezekowitz JA, Cheng MP, Ambrosy AP, Zannad F, Brophy JM, Giannetti N, Bessissow A, Kronfli N, Marelli A, Aziz H, Alqahtani M, Aflaki M, Craig M, Lopes RD, Ferreira JP. A randomized controlled trial of renin-angiotensin-aldosterone system inhibitor management in patients admitted in hospital with COVID-19. Am Heart J. 2022 May;247:76-89. doi: 10.1016/j.ahj.2022.01.015. Epub 2022 Feb 7. PMID 35143744
- [Derived] Aflaki M, Flannery A, Ferreira JP, Cheng MP, Kronfli N, Marelli A, Zannad F, Brophy J, Afillalo J, Huynh T, Giannetti N, Bessissow A, Ezekowitz JA, Lopes RD, Ambrosy AP, Craig M, Sharma A. Management of Renin-Angiotensin-Aldosterone System blockade in patients admitted to hospital with confirmed coronavirus disease (COVID-19) infection (The McGill RAAS-COVID- 19): A structured summary of a study protocol for a randomized controlled trial. Trials. 2021 Feb 5;22(1):115. doi: 10.1186/s13063-021-05080-4. PMID 33546734
- See also: The novel coronavirus 2019 (2019-nCoV) uses the SARS-coronavirus receptor ACE2 and the cellular protease TMPRSS2 for entry into target cells — https://www.biorxiv.org/content/10.1101/2020.01.31.929042v1
- See also: Power and sample size estimation for nonparametric composite endpoints: Practical implementation using data simulations. — https://digitalcommons.wayne.edu/cgi/viewcontent.cgi?article=2451&context=jmasm